CLINICAL TRIAL: NCT04578002
Title: Telestroke 2: Prehospital Triage of Patients With Suspected Stroke Using Onsite Mobile Telemedicine- Efficacy Study
Brief Title: Telestroke 2: Prehospital Triage of Patients With Suspected Stroke Using Onsite Mobile Telemedicine
Acronym: Telestroke 2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: propatient Forschungsstiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-0126; me20Lyrer
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Acute
Keywords: pre-hospital triage; Stroke, suspected; Telemedicine; telemedical triage; Door-to-treatment-time
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prehospital telemedical triage — Prehospital Triage of Patients with Suspected Stroke Using Onsite Mobile Telemedicine approach (interactive video and audio streaming). In patients with suspected stroke, a prehospital patient evaluation by end-to-end encrypted real-time audio- and video streaming from the pre-hospital setting to an in-hospital stroke physician, located at the University hospital of Basel, is requested and initiated (telestroke-path). The process is supervised and evaluated by an in-hospital stroke physician in real-time. Patients considered having an acute stroke will be directly transferred to cerebral imaging via CT. All other patients will follow conventional stroke path.

SUMMARY:
This study is to investigate clinical efficacy of the pre-hospital triage of patients with suspected acute stroke by using advanced telecommunication tools with digital audio and video real-time streaming.

DETAILED DESCRIPTION:
One of today's main challenges in stroke medicine is to further decrease event-to-treatment-time. On-site, pre-hospital, clinical assessment of patients with suspected acute stroke can optimize further diagnostic and treatment pathways after patient arrival at the dedicated stroke center. A telemedical approach (interactive video and audio streaming) allows time efficient pre-hospital triage, via patient evaluation by simple, pre-defined assessment measures and a standardized questionnaire. This study is to investigate clinical efficacy of the pre-hospital triage of patients with suspected acute stroke by using advanced telecommunication tools with digital audio and video real-time streaming.

ELIGIBILITY:
Inclusion Criteria:

* suspected acute stroke as per the first judgement of the paramedics on-site

Exclusion Criteria:

* Patients with a known history of epilepsia or non-epileptic seizures
* Patients after/while displaying an epileptic seizure
* Recent head trauma
* Patient with a reduced Glasgow Coma Scale or other condition not allowing Rapid Arterial oCclusion Evaluation (RACE) examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient aged ≥ 18 years with suspected acute stroke as per the first judgement of the paramedics on-site at the University hospital of Basel.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Door-to-treatment-time (minutes) | one point assessment at baseline
  Door-to-treatment-time (minutes), assessed as door-to-needle-time and door-to-groin-puncture-time.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) at 24hours | one point assessment at 24hours after hospital admission
  Score to quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
National Institutes of Health Stroke Scale (NIHSS) at 90 days | one point assessment at 90 days after hospital admission
  Score to quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
modified Rankin Scale (mRS) at 90 days | one point assessment at 90 days after hospital admission
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lyrer, Prof. Dr. med., Principal Investigator — Stroke Center, Neurology, University Hospital Basel
Locations (1):
- Stroke Center, Neurology, University Hospital Basel, Basel, Switzerland